CLINICAL TRIAL: NCT02005393
Title: A Concurrence Study of Diagnostic Visualization Comparing Flexible Spectral-Imaging Color Enhancement (FICE) With Olympus Narrow Band Imaging (NBI)
Brief Title: Study Comparing Flexible Spectral-Imaging Color Enhancement (FICE) With Olympus Narrow Band Imaging (NBI)
Acronym: FICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P-13-003
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Routine Endoscopy
Keywords: FICE; NBI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FICE Imaging System followed by NBI (Other): Images Captured with FICE Image Acquisition System (experimental) followed by NBI Image Acquisition System (standard of care); always in that order. Imaging took place in esophagus, gastric, duodenum and/or colon.
  Interventions: Device: FICE Image Acquisition followed by NBI Image Acquisition

INTERVENTIONS:
Device: FICE Image Acquisition followed by NBI Image Acquisition — Images Captured with FICE Device, followed by same locations imaged with NBI Image Acquisition System

SUMMARY:
The study is intended to test the image quality of the FICE system to the predicate device, Narrow Band Imaging (NBI). The hypothesis is the images are of equal quality.

DETAILED DESCRIPTION:
No additional description required.

ELIGIBILITY:
Inclusion Criteria:

* Referred for diagnostic endoscopy or colonoscopy
* Ability to comply and willingness to partake in study

Exclusion Criteria:

* less than 21 years of age
* is an inmate

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Moore, Study Director — FujiFilm Medical Systems USA
Locations (1):
- Mayo Clinic, Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty subjects were recruited at Mayo Clinic, Scottsdale between 23Oct2013 and 08Nov2013 to have two endoscopies completed - one using Fujifilm's endoscope and processor equipped with FICE, and the second immediately following with Olympus' endoscope and processor equipped with NBI.
Groups:
- FICE Image Acquisition Followed by NBI Image Acquisition: Images Captured with FICE Image Acquisition immediately followed by NBI Image Acquisition
  FICE Image Acquisition System: Images Captured with FICE Device
Period: Overall Study
Arm/Group | FICE Image Acquisition Followed by NBI Image Acquisition
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- FICE Image Acquisition Followed by NBI Image Acquisition: Images Captured with FICE Image Acquisition System immediately followed by Image Acquisition with NBI
  FICE Image Acquisition System: Images Captured with FICE Device
Arm/Group | FICE Image Acquisition Followed by NBI Image Acquisition
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Image Quality Scores Using Likert Scale
Description: Likert score ratings of image quality for FICE and NBI images. Each FICE setting was compared to NBI, to determine which FICE settings were equivalent to NBI.
  Likert Scores:
  1. Not seen;
  2. poor but usable, characteristic features are detectable but details are not fully reproduced; features just visible;
  3. good; allows an adequate assessment, details of anatomical structures are visible but not necessarily clearly defined; details emerging;
  4. very good; allows an excellent assesssment, anatomical details are clearly defined; details clear
Time Frame: One day
Population: All patients had imaging done with both FICE, immediately followed by NBI. Images for one subject were not included in the Reader Study due to an error on the Compact Flash card which resulted in three (3) corrupt FICE images (FICE settings 0, 1 & 2); therefore making 19 out of 20 participants analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FICE Image Acquisition Followed by NBI Image Acquisition: Images Captured with FICE Image Acquisition System, immediately followed by NBI Image Acquisition; always in that order.
  FICE Image Acquisition System: Images Captured with FICE Device
Arm/Group | FICE Image Acquisition Followed by NBI Image Acquisition
Number analyzed (Participants) | 19
units on a scale
  FICE 0 | 3.2 (0.7)
  FICE 1 | 3.3 (0.7)
  FICE 2 | 3.4 (0.6)
  FICE 3 | 3.3 (0.7)
  FICE 4 | 3.3 (0.8)
  FICE 5 | 3.1 (0.8)
  FICE 6 | 3.4 (0.7)
  FICE 7 | 3.0 (0.8)
  FICE 8 | 3.1 (0.7)
  FICE 9 | 3.2 (0.8)
  NBI | 3.1 (1.1)
Statistical Analysis 1: Comparison: FICE Image Acquisition Followed by NBI Image Acquisition; All 20 subjects enrolled in the study, including Subject 219 that was dropped from the Reader assessments due to corrupted images, were all rated as having similar white light images between the FICE and NBI procedures for each location used in the concurrence study. This assessment was intended to assure that no procedural sequence or visualization bias was introduced into the image acquisition process. The overall Reader mean (SD) for both FICE and NBI were equal to or greater than 3.0 (0.8); Test type: Non-Inferiority or Equivalence — Image settings were considered non-inferior if scores overlapped within 1 SD of mean; The results reported utilized the average Likert scores for each of the 3 readers, for each of the FICE settings (0-9), as compared to FICE. The overall Reader mean (SD) for both FICE and NBI were equal to or greater than 3.0 (0.8).The overall mean scores were comparable between FICE and NBI to provide acceptable diagnostic image visualization quality

ADVERSE EVENTS:
Time Frame: There were no AE's for this study, however an event would have been considered an AE from the time they started the procedure, until the patient life the hospital for the day.
Description: No AE's (or SAE's) reported.
Groups:
- FICE Image Acquisition Followed by NBI Image Acquisition: Images Captured with FICE Image Acquisition System, immediately followed by Image Acquisition with NBI
  FICE Image Acquisition System: Images Captured with FICE Device
  No AE's
Arm/Group | FICE Image Acquisition Followed by NBI Image Acquisition
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less